CLINICAL TRIAL: NCT03159078
Title: Polymyxin B Monotherapy Versus Polymyxin B-Carbapenem Combination Therapy in Critically Ill Patients With Multi-drug Resistant Gram-negative Infection: A Prospective, Parallel-Group, Double-Blind, Randomized Controlled Study
Brief Title: Polymyxin B Monotherapy vs Combination Therapy in Critically Ill Patients With Multi-drug Resistant Pathogens
Acronym: MUSEUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1210116
Record Dates: First submitted 2017-05-10; First posted 2017-05-18 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Trauma; Resistant Infection; Critical Illness
Keywords: Acinetobacter; Polymyxins; Imipenem; Pseudomona; Klebsiella
MeSH Terms: conditions — Wounds and Injuries; Critical Illness; Pseudomonas Infections; Klebsiella Infections | interventions — Polymyxin B; Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Intervention Model Description: One arm with Polyxyxin B monotherapy and another arm with Polymyxin B plus carbapenem
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind, Double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Polymyxin B monotherapy (Other): Intravenous piggyback with Polymyxin B and control(Normal saline)
  Interventions: Drug: Polymyxin B
- Polymyxin B plus Carbapenem (Experimental): Intravenous piggyback with Polymyxin B plus Carbapenem
  Interventions: Drug: Polymyxin B

INTERVENTIONS:
Drug: Polymyxin B — Comparison of Poly B monotherapy vs Polymyxin B plus carbapenem in MDR infections
  Other Names: Imipenem, (Primaxin)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of polymyxin B as monotherapy versus a combined polymyxin B-carbapenem therapy against multidrug-resistant (MDR) gram negative infections. The investigators intend to evaluate if this synergistic drug regimen correlates with improved outcomes against gram-negative infections in critically ill patients including: better clinical resolution, reduced length of stay at hospital, reduced length of stay at the intensive care unit, and less recurrence of infection.

DETAILED DESCRIPTION:
The "MUSEUM" trial is a single-center, prospective, parallel-group, double-blind, randomized, controlled study design. The trial will be conducted at the Intensive Care Unit of the Puerto Rico Trauma Hospital located in San Juan, Puerto Rico. Patients with clinical and microbiological evidence of an Multi-drug resistant infection related to Hospital-acquired pneumonia (HAP), Ventilator-associated pneumonia (VAP), Complicated Urinary tract infection (cUTI) or Bloodstream infection (BSI) will be considered candidates for the study. The pathogen should be resistant to all antibiotics except to polymyxin B. With a predicted survival rate of 67% (hazard ratio of 0.33), a significance of α = 0.05, power of 80%, and assuming a dropout rate of 15%, the estimated sample size is n = 40 patients (20 per group). In terms of safety, the most clinically relevant adverse effects are nephrotoxicity and neurotoxicity, which will be evaluated and adjudicated. The recurrence of infection will be defined as a new superinfection by the same or other species than the initial infection that is multidrug-resistant. Length of stay at the Hospital will be measured from the day of admission until the day of discharge. Length of stay in the ICU will be measured from the day of admission until the day of discharge from the unit. To our knowledge, this will be the first prospective, double blind, randomized, controlled clinical trial in representation of the critically ill trauma patients infected with Multi-drug resistant pathogens.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older admitted to the Intensive Care Unit of the Puerto Rico Trauma Hospital ° Consent form signed,
* Clinical and microbiological evidence of a MDR infection related to HAP, VAP, cUTI or BSI.
* The pathogen should be resistant to almost all antibiotics, AND/OR intermediate resistant to some of the antibiotics, AND/OR susceptible only to a class of antibiotic (i.e. aminoglycosides which are NOT recommended as monotherapy), AND/OR the clinician decision is to start the patient on polymyxin B due to severity of the infection.
* Patient with a diagnosis of MDR infection, who have not received antibiotics at all; OR if received would be < 72 hours with polymyxin B or imipenem at/or after the diagnosis of MDR AND/OR at the time of randomization
* Have a life expectancy of > 24 hours according to the attending physician's criteria.

Exclusion Criteria:

* Pregnant woman
* Prisoners
* Severe hepatic failure (defined by serum conjugated bilirubin > 3 mg/dL)
* End-stage renal disease requiring hemodialysis
* Hypersensitivity to any study drug
* Septic shock at the moment of randomization
* Died within 48 hours of starting the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of the evidence of clinical infection | 7-14 days, according to site of infection
  Resolution of infection will be subjective to clinical criteria of the physician, AND patient has to be afebrile (temperature < 38°C), or normothermic (temperature 36-37.5°C), AND have white blood cell count within normal limits (> 4,000 and < 10,000 cells/mm3).

SECONDARY OUTCOMES:
30-day mortality | 30 days
  Thirty-day (30-day) mortality will be measured from the day of hospital admission until discharge.
Recurrence of infection | 30 days
  The recurrence of infection will be defined as a new superinfection by the same or other species than the initial infection that is multidrug-resistant.
Length of stay at Hospital | 30 days
  Will be measured from the day of hospital admission until discharge.
Length of stay at ICU. | 30 days
  Will be measured from the day of ICU admission until transfer or discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Maldonado Lozada, PharmD, Principal Investigator — School of Pharmacy, University of Puerto Rico
Locations (1):
- Trauma Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Struelens MJ. The epidemiology of antimicrobial resistance in hospital acquired infections: problems and possible solutions. BMJ. 1998 Sep 5;317(7159):652-4. doi: 10.1136/bmj.317.7159.652. No abstract available. PMID 9727997
- [Result] Sandri AM, Landersdorfer CB, Jacob J, Boniatti MM, Dalarosa MG, Falci DR, Behle TF, Bordinhao RC, Wang J, Forrest A, Nation RL, Li J, Zavascki AP. Population pharmacokinetics of intravenous polymyxin B in critically ill patients: implications for selection of dosage regimens. Clin Infect Dis. 2013 Aug;57(4):524-31. doi: 10.1093/cid/cit334. Epub 2013 May 22. PMID 23697744
- [Result] Zavascki AP, Bulitta JB, Landersdorfer CB. Combination therapy for carbapenem-resistant Gram-negative bacteria. Expert Rev Anti Infect Ther. 2013 Dec;11(12):1333-53. doi: 10.1586/14787210.2013.845523. Epub 2013 Nov 6. PMID 24191943
- [Result] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Result] Landman D, Georgescu C, Martin DA, Quale J. Polymyxins revisited. Clin Microbiol Rev. 2008 Jul;21(3):449-65. doi: 10.1128/CMR.00006-08. PMID 18625681
- [Result] Kassamali Z, Jain R, Danziger LH. An update on the arsenal for multidrug-resistant Acinetobacter infections: polymyxin antibiotics. Int J Infect Dis. 2015 Jan;30:125-32. doi: 10.1016/j.ijid.2014.10.014. Epub 2014 Nov 5. PMID 25461655
- [Result] Falagas ME, Rafailidis PI, Kasiakou SK, Hatzopoulou P, Michalopoulos A. Effectiveness and nephrotoxicity of colistin monotherapy vs. colistin-meropenem combination therapy for multidrug-resistant Gram-negative bacterial infections. Clin Microbiol Infect. 2006 Dec;12(12):1227-30. doi: 10.1111/j.1469-0691.2006.01559.x. PMID 17121631
- [Result] Rigatto MH, Vieira FJ, Antochevis LC, Behle TF, Lopes NT, Zavascki AP. Polymyxin B in Combination with Antimicrobials Lacking In Vitro Activity versus Polymyxin B in Monotherapy in Critically Ill Patients with Acinetobacter baumannii or Pseudomonas aeruginosa Infections. Antimicrob Agents Chemother. 2015 Oct;59(10):6575-80. doi: 10.1128/AAC.00494-15. Epub 2015 Aug 10. PMID 26259799
- [Result] Daikos GL, Tsaousi S, Tzouvelekis LS, Anyfantis I, Psichogiou M, Argyropoulou A, Stefanou I, Sypsa V, Miriagou V, Nepka M, Georgiadou S, Markogiannakis A, Goukos D, Skoutelis A. Carbapenemase-producing Klebsiella pneumoniae bloodstream infections: lowering mortality by antibiotic combination schemes and the role of carbapenems. Antimicrob Agents Chemother. 2014;58(4):2322-8. doi: 10.1128/AAC.02166-13. Epub 2014 Feb 10. PMID 24514083
- [Result] Tumbarello M, Viale P, Viscoli C, Trecarichi EM, Tumietto F, Marchese A, Spanu T, Ambretti S, Ginocchio F, Cristini F, Losito AR, Tedeschi S, Cauda R, Bassetti M. Predictors of mortality in bloodstream infections caused by Klebsiella pneumoniae carbapenemase-producing K. pneumoniae: importance of combination therapy. Clin Infect Dis. 2012 Oct;55(7):943-50. doi: 10.1093/cid/cis588. Epub 2012 Jul 2. PMID 22752516
- [Result] Sobieszczyk ME, Furuya EY, Hay CM, Pancholi P, Della-Latta P, Hammer SM, Kubin CJ. Combination therapy with polymyxin B for the treatment of multidrug-resistant Gram-negative respiratory tract infections. J Antimicrob Chemother. 2004 Aug;54(2):566-9. doi: 10.1093/jac/dkh369. Epub 2004 Jul 21. PMID 15269195
- [Result] Anthony KB, Fishman NO, Linkin DR, Gasink LB, Edelstein PH, Lautenbach E. Clinical and microbiological outcomes of serious infections with multidrug-resistant gram-negative organisms treated with tigecycline. Clin Infect Dis. 2008 Feb 15;46(4):567-70. doi: 10.1086/526775. PMID 18199038
- [Result] Qureshi ZA, Paterson DL, Potoski BA, Kilayko MC, Sandovsky G, Sordillo E, Polsky B, Adams-Haduch JM, Doi Y. Treatment outcome of bacteremia due to KPC-producing Klebsiella pneumoniae: superiority of combination antimicrobial regimens. Antimicrob Agents Chemother. 2012 Apr;56(4):2108-13. doi: 10.1128/AAC.06268-11. Epub 2012 Jan 17. PMID 22252816
- [Result] Maragakis LL, Perl TM. Acinetobacter baumannii: epidemiology, antimicrobial resistance, and treatment options. Clin Infect Dis. 2008 Apr 15;46(8):1254-63. doi: 10.1086/529198. PMID 18444865
- [Result] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Result] Seifert H. The clinical importance of microbiological findings in the diagnosis and management of bloodstream infections. Clin Infect Dis. 2009 May 15;48 Suppl 4:S238-45. doi: 10.1086/598188. PMID 19374579
- [Result] Durante-Mangoni E, Signoriello G, Andini R, Mattei A, De Cristoforo M, Murino P, Bassetti M, Malacarne P, Petrosillo N, Galdieri N, Mocavero P, Corcione A, Viscoli C, Zarrilli R, Gallo C, Utili R. Colistin and rifampicin compared with colistin alone for the treatment of serious infections due to extensively drug-resistant Acinetobacter baumannii: a multicenter, randomized clinical trial. Clin Infect Dis. 2013 Aug;57(3):349-58. doi: 10.1093/cid/cit253. Epub 2013 Apr 24. PMID 23616495
- [Result] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Result] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Result] Michel DJ, Knodel LC. Comparison of three algorithms used to evaluate adverse drug reactions. Am J Hosp Pharm. 1986 Jul;43(7):1709-14. PMID 3752106
- [Result] Siddiqui NU, Qamar FN, Jurair H, Haque A. Multi-drug resistant gram negative infections and use of intravenous polymyxin B in critically ill children of developing country: retrospective cohort study. BMC Infect Dis. 2014 Nov 28;14:626. doi: 10.1186/s12879-014-0626-9. PMID 25430979
- See also: Trial for the Treatment of Extensively Drug-Resistant Gram-negative Bacilli — https://clinicaltrials.gov/ct2/show/record/nct01597973?term=nct01597973&rank=1
- See also: Multicenter Open-label Randomized Controlled Trial (RCT) to Compare Colistin Alone Versus Colistin Plus Meropenem — https://clinicaltrials.gov/ct2/show/record/nct01732250?term=nct01732250&rank=1
- See also: Primaxin I.V. (Imipenem and Cilastatin for IV Injection). — https://www.merck.com/product/usa/pi_circulars/p/primaxin/primaxin_iv_pi.pdf